CLINICAL TRIAL: NCT05148000
Title: Open-label Study to Assess Aesthetic Improvement Following Treatment With QM1114-DP in Subjects With Moderate to Severe Lateral Canthal Lines and Glabellar Lines
Brief Title: Assess Aesthetic Improvement With QM1114-DP in Subjects With Moderate to Severe Lateral Canthal Lines and Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43QM2107
Record Dates: First submitted 2021-10-31; First posted 2021-12-07 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-02

CONDITIONS: Glabellar Frown Lines; Canthal Lines

STUDY DESIGN:
Intervention Model Description: Open Label single site study for treatment of GL and LCL with single treatment of QM1114-DP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QM1114-DP (Experimental): QM1114-DP
  Interventions: Biological: QM1114-DP

INTERVENTIONS:
Biological: QM1114-DP — QM1114-DP

SUMMARY:
This study to assess aesthetic improvement following treatment with QM1114-DP.

DETAILED DESCRIPTION:
This is an open-label, single-center multi-center study to assess aesthetic improvement in the Glabellar and Lateral Canthal regions following treatment with QM1114-DP.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years or older
* Moderate to severe bilaterally symmetrical LCL as assessed by the investigator
* Moderate to severe GL at maximum frown as assessed by the Investigator

Exclusion Criteria:

* Previous use of any botulinum toxin in facial areas within 9 months prior to study treatment
* Female who is pregnant, breast feeding or intends to conceive a child during the study.
* Known allergy to hypersensitivity or any component of the Investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Responders in QM1114-DP versus Placebo using the Global Aesthetic Improvement Scale (GAIS) at maximum frown at Month 1 | 1 month
  Responder Rate is defined as a subject who responds at least Improved on the GAIS at maximum frown
Responders in QM1114-DP versus Placebo using the Global Aesthetic Improvement Scale (GAIS) at maximum smile at Month 1 | 1 month
  Responder Rate is defined as a subject who responds at least Improved on the GAIS at maximum smile

CONTACTS AND LOCATIONS:
Locations (1):
- Galderma Research Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No